CLINICAL TRIAL: NCT01557868
Title: Prediction of Response to Intra-articular Injections of Hyaluronic Acid for Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Orthopaedic Society for Sports Medicine (Other)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AOSSM 51H
Record Dates: First submitted 2012-03-12; First posted 2012-03-20 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synvisc (hylan G-F 20) (Active Comparator)
  Interventions: Device: hylan G-F 20
- Euflexxa (1% sodium hyaluronate) (Active Comparator)
  Interventions: Device: 1% sodium hyaluronate

INTERVENTIONS:
Device: hylan G-F 20 — Three 2 cc injections at weekly intervals
  Other Names: Synvisc
  Arms: Synvisc (hylan G-F 20)
Device: 1% sodium hyaluronate — Three 2 cc injections at weekly intervals
  Other Names: Euflexxa
  Arms: Euflexxa (1% sodium hyaluronate)

SUMMARY:
The purpose of this study is to evaluate whether the investigators can develop a computer algorithm to predict which individual patients will respond to injections of hyaluronic acid (HA) products for knee osteoarthritis.

DETAILED DESCRIPTION:
Background Osteoarthritis (OA) of the knee is a debilitating condition that affects an estimated 21 million Americans. This number is expected to rise steadily as the population ages. The medical expenditures associated with arthritis and other rheumatic conditions in the United States have increased from $50 billion in 1997 to $86 billion in 2003. In 2003, almost 420,000 total knee replacements were performed, primarily for arthritis. Injections of hyaluronic acid (HA) have been shown to provide symptom relief for many OA patients who have failed to respond to conservative interventions. Many other patients, however, experience only slight or no improvement. The results from this study will allow physicians to identify whether a patient is likely or not likely to respond well to HA therapy leading to improved treatment success rates.

Goals This study has two related goals: 1) to identify patient and treatment factors that predict response to intra-articular injections of hyaluronic acid for knee osteoarthritis using multivariable analysis and 2) develop mathematical and statistical models that will predict individual patient response to HA for knee OA.

It is anticipated that the investigators will develop computer software in this study that can support clinical decision making related to viscosupplementation in the treatment of knee OA. If this project yields successful patient predictive models, physicians who are considering a trial of HA for a patient will have some empirical basis for treatment selection. Eventually a physician would be able to assess a relatively small number of variables for a patient and then be provided with predictions regarding treatment response.

**Please note that the study site at the Naval Medical Center in Portsmouth, Virginia can only enroll patients who are eligible to be treated at a military facility.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee osteoarthritis presenting to physician's office
* Radiographic evidence of knee osteoarthritis
* Age 18 years or older
* Failed minimum of 3 months of non-operative treatment, including, but not limited to, Tylenol, anti-inflammatory medication, cortisone injection, physical therapy, bracing, and/or heel wedge
* Symptoms for at least 3 months

Exclusion Criteria:

* Associated ligamentous instability
* History of deep knee infection
* Candidate for total knee arthroplasty or arthroscopy
* Peripheral neuropathy.
* X-rays that are completely negative and only MRI evidence or arthroscopic evidence (from previous arthroscopy) of OA.
* Prior HA injections at any point in the past
* Chondrocalcinosis
* Patients with precautions or contraindications for viscosupplementation use
* Cortisone injection within past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Marx, MD, Study Chair — Hospital for Special Surgery, New York; Marlene DeMaio, MD, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Naval Medical Center Portsmouth (this site can only enroll patients who are eligible to be treated at a military facility), Portsmouth, Virginia, United States

REFERENCES:
- See also: Information on Osteoarthritis from the National Institutes of Health — http://www.niams.nih.gov/Health_Info/Osteoarthritis/default.asp
- See also: Cochrane Review Article Abstract on Viscosupplementation for Knee Osteoarthritis — http://www.ncbi.nlm.nih.gov/pubmed/16625635

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synvisc (Hylan G-F 20) | Euflexxa (1% Sodium Hyaluronate)
Started | 103 | 95
Completed | 76 | 65
Not Completed | 27 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synvisc (Hylan G-F 20) | Euflexxa (1% Sodium Hyaluronate) | Total
Number analyzed (Participants) | 103 | 95 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (9.6) | 43.3 (10.4) | 45.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 35 | 78
  Male | 60 | 60 | 120
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 5 | 6
  Black/African American | 33 | 21 | 54
  Hispanic | 5 | 6 | 11
  White | 62 | 62 | 124
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 103 | 95 | 198

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Scale
Description: The KOOS is 42-item patient-report questionnaire that assesses symptoms and problems associated with knee injury and osteoarthritis. It yields scores for five scales including Pain, Other Symptoms, Function in Daily Living, Function in Sport/Recreation, and Knee-Related Quality of Life. We used only the Pain scale which has a range of 0 to 100 where 100 represents the "best" score, i.e., no pain. We reported differences in baseline Pain scale score from Pain scale score at 6 months so these scores could theoretically range from -100 (moving from no pain to maximum pain) to 100 (moving from maximum pain to no pain). Positive change scores represent improvement from baseline.
Time Frame: Baseline and at 6 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc (Hylan G-F 20) | Euflexxa (1% Sodium Hyaluronate)
Number analyzed (Participants) | 76 | 65
units on a scale | 12.8 (18.9) | 9.8 (20.5)

2. Secondary Outcome: Visual Analogue Scale (VAS) at 6 Months
Description: The VAS is a patient-reported assessment of knee pain. Patients mark on a line (0-100mm) their current level of knee pain while moving where 0 represent no pain and 100 represents maximum pain. We report changes in VAS pain rating between baseline and 6 month follow-up. Therefore scores can theoretically range from -100 (moving from maximum pain to no pain) to 100 (moving from no pain to maximum pain). Negative change scores represent decreases in perceived pain or improvement.
Time Frame: Assessments were at baseline to 6 month follow-up
Population: The discrepancy between the number of subjects included in this analysis (140) and the number of subjects reported completing the study (141) is due to a missing values for one subject for this variable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc (Hylan G-F 20) | Euflexxa (1% Sodium Hyaluronate)
Number analyzed (Participants) | 76 | 64
units on a scale | -13.7 (28.4) | -10.7 (25.4)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Synvisc (Hylan G-F 20) | Euflexxa (1% Sodium Hyaluronate)
Serious Adverse Events (participants affected / at risk) | 8/103 | 1/95
Other Adverse Events (participants affected / at risk) | 0/103 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synvisc (Hylan G-F 20) (N=103) | Euflexxa (1% Sodium Hyaluronate) (N=95)
Knee Effusion (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No